CLINICAL TRIAL: NCT06652594
Title: Effect of "eye" Education for Parents on Myopia Prevention and Control in Children
Brief Title: "Eye" Education for Parents and Myopia Control in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Shi-Ming Li, Professor, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-2G-1081
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Children; Health Education; Anxiety
MeSH Terms: conditions — Health Education; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eye Education Intervention (Experimental): Doctors and nurses will educate parents about eye health in response to their child's myopia progression at baseline, 1 month, 3 months, 6 months.
  Interventions: Behavioral: Eye Education Intervention
- Control (Experimental): Parents in the control group will not receive eye health education information from doctors and nurses.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Eye Education Intervention — Doctors and nurses will educate parents about eye health in response to theirchild's myopia progression at baseline, 1 month, 3 months, 6 months.
  Arms: Eye Education Intervention
Behavioral: Control — Parents in the control group will not receive eye health education informationfrom doctors and nurses.
  Arms: Control

SUMMARY:
This is a randomized controlled trial aimed to explore the effect of behavioral interventions based on doctors' and nurses' health education on the onset and development of myopia in children's. Participants were randomly assigned to one of two groups: eye health intervention, or the control group. Intervention group's parents would reveive eye health education in response to their children's myopia progression at baseline, 1 month, 3 months, and 6 months, while the control group did not receive any. Visual acuity, cycloplegic refraction, axial length, Strengths and Difficulties Questionnaire, and Generalized Anxiety Disorder 7-item Scale were the main outcomes and measures.

DETAILED DESCRIPTION:
After doctors' and nurses' education, parents would keep a diary to regulate the children's "Sedentary", "Sunshine", "Sleep", "Screen", and "Stress" that is, the "5S" eye education. To urging parents pay attention to the children's eye behavior every day, and targeted to children "eye" education to delay the occurrence and development of myopia and reduce the incidence of high myopia.

ELIGIBILITY:
Inclusion Criteria

1. Children aged 5-17;
2. Removing flexible lenses for at least 1 week, flexible astigmatism and hard lenses for at least 3 weeks, orthokeratology lenses for at least 3 months;
3. Best corrected visual acuity of either eye were all ≥ 1.0;
4. The range of myopia in either eye was -15 D ≤ SE ≤ +2.0 D;
5. Astigmatism of either eye less than -5.0 D;
6. Anisometropia ≤ -1.5 D;
7. There was no active ocular inflammatory diseases; no obvious corneal cloud or macula, anormal corneal topography, and no tendency of keratoconus.
8. Intraocular pressure of either eye is of 10 to 21 mmHg;
9. On the basis of full understanding, children and their guardians sign the informed consent;

Exclusion Criteria:

1. Amblyopia: best corrected visual acuity (BCVA) of either eye less than 1.0 for children over 6 years old;
2. Active ocular inflammatory diseases, such as uveitis and other inflammatory diseases;
3. Secondary myopia, genetic disease or connective tissue- related myopia;
4. Moderate or severe ptosis;
5. Congenital cataract, glaucoma;
6. Other fundus diseases other than myopic related fundus lesions;
7. Intraocular or refractive surgery history;
8. The refractive medium is turbid, and it is impossible to take a clear fundus image; (9)Unable to cooperate with fundus image shooting and other examination;

(10)Do not receive cycloplegia or have contraindications; (11)Poor overall condition, unable to follow up for a long time; (12)The subject refuses to participate in the research; (13)Other cases in which the researcher judges that it is not suitable for participation in the study.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 498 (Estimated)
Dates: Start 2024-10-19 (Estimated); Primary Completion 2025-04-19 (Estimated); Study Completion 2025-04-19 (Estimated)

PRIMARY OUTCOMES:
Axial Length | Baseline, 1 month, 3 months, 6 months.
  Ocular biometry was used for measuring the axial length, which is the physical distance between the anterior corneal pole and the retinal structure at the posterior pole.
Cycloplegic Refraction | Baseline, 1 month, 3 months, 6 months.
  Cycloplegic refractive errors were measured with an autorefractor.

SECONDARY OUTCOMES:
Visual acuity | Baseline, 1 month, 3 months, 6 months.
  The visual acuity of the children is assessed through a self-administered vision test conducted by their guardians via WeChat mini program.
Anxiety Disorder Screening 7-item Scale | Baseline, 6 month
  Assessing changes in parents' anxiety before and after the intervention.
Strengths and Difficulties Questionnaire | Baseline, 6 month.
  Assessing changes in parent-child relationships before and after the intervention.

OTHER OUTCOMES:
Fundus Image | Baseline, 1 month, 3 months, 6 months.
  Two fundus photographs were taken for each subject, centered on the optic disc and macula with a 45° field of view. If the quality of the photographs was low, they were retaken.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No